"Evaluation of The Effect of Neck and Trunk Stabilization Exercises on Quality of Life and Communication in Children with Cerebral Palsy with Oral Motor Problem"

NCT04214080

23.03.2018

## **Informed Consent Form**

I would like to do a research called "Evaluation of the Effect of Neck and Trunk Stabilization Exercises on Quality of Life and Communication in Children with Cerebral Palsy with Oral Motor Problem". In this research, your child's communication and quality of life will be evaluated. The research will be performed under the direction of Assoc. Dr. Aysel YILDIZ OZER, and Pt. Nasim EJRAEI from Marmara University Health Sciences Institute, Department of Physiotherapy and Rehabilitation, Department of Physiotherapy and Rehabilitation.

You are invited to a study. It is very important to understand why and how to do the research before making a decision. Please take some time and carefully read the information below, discuss with others if you wish. If there is an unclear section or if you need more detailed information, you can get information from us. You are invited to our research because you meet the criteria for inclusion in the research sought by the participants. There was a relationship between vocal functions and posture, active trunk movements has an important role in sound production and lastly trunk stabilization, balance and activity level components are in relationship with each other. Thus in this study, it was aimed to investigate the effects of neck and trunk stabilization exercises on communication, activities of daily living and quality of life in children with CP with oral motor problem. Children who volunteer to participate in this study will receive eating training in addition to the physiotherapy program applied based on the principles the Neurodevelopmental Treatment and will receive therapy that includes trunk exercises based on the principles of Neurodevelopmental Treatment. Both types of therapy programs do not harm your child without any especial risks. The evaluations applied to the participants participating in our research have no known harm. If you are harmed in any way from the evaluations, the necessary applications will be met by the researchers without any response. Before and after this exercise program, your child will be evaluated.

We would like to state that participation is voluntary and refusal to participate will not lead to any punishment or loss of any benefit. Likewise, after you agree to participate in the research, you can withdraw from the research without showing any reason anywhere in the research. No fees will be charged for this, neither from you nor from your Social Security. Although it may be beneficial for you to participate in the research immediately, it is hoped that our research results will benefit the institution, society or science in the future.

I have read the entire information form clearly or understandably read/translated to me

as I do not know the language/reading. I was given the opportunity to ask, evaluate and make

decisions about my health status both during and after my application and while filling out this

form. All treatment and diagnostic alternatives, including the possibility of non-treatment, and

whether there are risks and dangers were explained.

Name-Surname of the participant and his/her legal representative:

**Date/Signature:** 

I gave the patient the necessary information about the disease and the procedures to be

applied. I believe that the patient understands this information, asks me the questions he wants

to ask, and accepts the process with his free will.

Researcher: Pt. Nasim EJRAEI

Address: Marmara University Başıbüyük Health Campus, Health Sciences Institute

Directorate, Başıbüyük Yolu 9/3 34854 Başıbüyük / Maltepe / Istanbul

**Telephone:** 0539 298 71 26

**E-mail:** ejraeinasim@yahoo.com

**Date/Signature:**